CLINICAL TRIAL: NCT01141140
Title: (Mis)Perceptions About Healthy Eating: Effects on Food Intake and Appetite in Men and Women
Acronym: COLLATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government); Danone Institute International (Other)
Responsible Party: Principal Investigator, Véronique Provencher, Professeur sous octroi, Laval University
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: INAF 2009-117
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Eating; Obesity
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- M-NO-NR (Other): Men (M) non-obese (NO) and non-restrained (NR).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy
- M-NO-R (Other): Men (M) non-obese (NO) and restrained (R).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy
- M-O-NR (Other): Men (M) overweight or obese (O) and non-restrained (NR).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy
- M-O-R (Other): Men (M) overweight or obese (O) and restrained (R).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy
- W-NO-NR (Other): Women (W) non-obese (NO) and non-restrained (NR).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy
- W-NO-R (Other): Women (W) non-obese (NO) and restrained (R).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy
- W-O-NR (Other): Women (W) overweight or obese (O) and non-restrained (NR).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy
- W-O-R (Other): Women (W) overweight or obese (O) and restrained (R).
  Interventions: Behavioral: Healthy; Behavioral: Diet; Behavioral: Unhealthy

INTERVENTIONS:
Behavioral: Healthy — Favourable nutritional characteristics.
Behavioral: Diet — Benefits of an ingredient/nutrient for weight management
Behavioral: Unhealthy — Hedonic characteristics and less healthy ingredients.

SUMMARY:
In the face of an increased prevalence of obesity and chronic diseases in Canada, much effort has been invested to educate the population about healthy eating. Although Canadians are now aware of the importance of healthier food habits, rates of obesity and chronic diseases are still increasing. In addition, even if different labelling strategies are used to identify healthier foods in the market, consumers remain confused about what healthy eating should be. Might describing foods as healthy have unintended side-effects on food intake? Previous literature has shown that perceptions about the healthiness of foods may bias estimations of caloric content of foods, leading consumers to underestimate the caloric content of "healthy" food choices. Indeed, the investigators have recently shown that perceiving a food as healthy increased intake of that food by 35% in undergraduate female students. The general objective of the proposed research is to investigate whether food perceptions influence intake and appetite sensations in normal-weight and overweight/obese restrained and unrestrained males and females. This laboratory study, in which perceived healthiness and "fatteningness" of oatmeal-raisin cookies will be manipulated during an ad libitum single-meal occasion, will increase the investigators knowledge of the effects of external cues (and other psychological and physiological factors) on the control of food intake. Because the popularity and demand for nutrition information is increasing, such information is needed to improve clinical practices aiming at promoting sustainable healthy eating habits to help individuals achieve and maintain a healthy weight.

DETAILED DESCRIPTION:
The laboratory study will be conducted at the Clinical Investigation Unit (CIU) of the Institute of Nutraceuticals and Functional Foods (INAF). Food-related variables (perceived healthiness and "fatteningness" of foods) will be manipulated during an ad libitum single-meal test. We will examine the effects of these variables on food intake and appetite sensations in male and female normal-weight and overweight/obese restrained and unrestrained eaters. Each participant will be tested on an individual basis, during a 2-hour experimental session (randomized sessions between 11:00 a.m. and 5:00 p.m.). Because participants might change their eating behaviors if they become aware of the true purpose of the study, deception must be used. Males and females will thus be recruited to participate in an ostensible market-research study involving a taste-rating task, and each participant will then be carefully debriefed at the end of the experiment.

Male and female normal-weight with a body mass index (BMI) ≥18.5kg/m2 and <25kg/m2 and overweight/obese with a BMI ≥25kg/m2, restrained and unrestrained eaters will be randomly assigned to one of three experimental conditions ("healthy," "diet," and "unhealthy"). A plate of about 1000 grams (g) of bite-sized oatmeal-raisin cookies will be presented to each participant. On average, one bite-size cookie is about 10g, which represents approximately 40 kilocalories (kcal) per cookie. The manipulation of healthiness and "fatteningness" perceptions of the oatmeal-raisin cookies will be performed verbally by the experimenter as follows. In the "healthy" condition, the description will emphasize nutritional characteristics (e.g., high in fibre, low in saturated fat and free from trans-fat), so the overall healthiness of the snack will be highlighted. In the "diet" condition, the description will emphasize the benefits of oatmeal fibre for weight management (e.g., helps to cope with hunger), thereby highlighting the weight-loss potential of the snack. In the "unhealthy" condition, the description will emphasize hedonic characteristics of the food and less healthy ingredients (e.g. gourmet cookies, contains butter and sugar), so some inherent unhealthy aspects of the snack will be highlighted.

Males and females involved in the study will be invited to participate in a market-research study investigating various dimensions of a new snack product. A telephone screening interview will first be conducted for all subjects interested in participating in the study to ensure that they meet our inclusion criteria, to facilitate randomization prior to the experiment session and to set the appointment with the participant. During this interview, each participant will be informed that this market-research study involves a taste-rating task in which they will taste and rate a new snack food. They will have to self-report their weight and height, and answer descriptive questions about inclusion criteria (e.g., history of health problems, current medications, liking of the tested food, and prior participation in studies). They will also have to complete the Restraint Scale to assess whether they exhibit behavioral and attitudinal concerns about dieting and weight control. Each participant will then be categorized as a restrained eater (≥12 in males and ≥15 in females) or unrestrained eater (<12 in males and <15 in females). Following the categorization established by the Restraint Scale and BMI calculation, each participant will then be randomly assigned to one of the experimental conditions, according to restraint and weight status (Note that randomization will be adjusted according to the measured BMI). The telephone screening interview will be conducted at least one week prior to the appointment at the CIU to ensure that having been asked about restraint and weight status will not affect participants' food intake and appetite sensations by making restraint and weight salient during the experiment. To standardize food intake and to insure that subjects have comparable baseline appetite sensations across experimental manipulations, participants will be asked to refrain from eating oatmeal-raisin cookies (tested food) for at least 24 hours prior to the experiment, and to arrive at the CIU for the appointment in a pre-meal state (i.e., at least 2 hours without food prior to the experiment). Because physical activity might have an impact on appetite sensations, participants will also be asked to refrain from doing any strenuous exercise at least for 24 hours before the experiment. Note that the experimenter in the study will strictly follow a detailed script when testing each participant to ensure that the testing will be consistent between all participants.

ELIGIBILITY:
Inclusion Criteria:

* Stable weight (± 2.5 kg) for at least 2 months prior to the study.
* Females will be tested in the follicular phase of their menstrual cycle to control for potential impact of hormonal variation on appetite measurements and food intake.

Exclusion Criteria:

* They will not be taking medication (e.g., corticosteroids, tricyclic antidepressants, atypical antipsychotics) and not present chronic health problems (e.g., eating disorders, diabetes, hyperthyroidism).
* No pregnant women nor lactating women.
* Aversion to the snack food used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Single-meal intake | 12-24-2010
  The amount of food eaten during the meal (grams and calories).

SECONDARY OUTCOMES:
Appetite sensations | 12-24-2010
  Visual-analogue ratings of desire to eat, hunger, fullness, and prospective food consumption (measured in millimeters).

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Provencher, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceuticals and Functionnal Foods (INAF), Québec, Quebec, Canada